CLINICAL TRIAL: NCT01653314
Title: A Randomized, Open-label, Single Dose, 2-Treatment, 2-Period, 2-Way Crossover Study to Assess Safety and Pharmacokinetics of Megavec 400 mg (Imatinib Mesylate) Under Fasted Conditions in Healthy Male Subjects
Brief Title: Megavec 400 mg (Imatinib Mesylate) in Healthy Adult Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: DW_MGV001
Record Dates: First submitted 2012-07-25; First posted 2012-07-31 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
MeSH Terms: interventions — Imatinib Mesylate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Megavec (Experimental)
  Interventions: Drug: Megavec; Drug: Glivec
- Glivec (Active Comparator)
  Interventions: Drug: Megavec; Drug: Glivec

INTERVENTIONS:
Drug: Megavec
Drug: Glivec

SUMMARY:
The purpose of this Study is to Assess Safety and Pharmacokinetics of megavec 400 mg (Imatinib mesylate) under Fasted Conditions in Healthy Male Subjects.

ELIGIBILITY:
* Inclusion Criteria:

  * Healthy and male subjects aged 20 to 55 years
  * The subject has a Body weight ≥55 kg and ideal body weight (IBW) within ±20%
  * A Subject who was judged to be healthy by the investigator to participate in this study based on screening results (according to standard reference index updated recently)
  * A subject who provided written informed consent to participate in this study and cooperative with regard to compliance with study related constraints.
* Exclusion Criteria:

  * A subject with sign or symptoms or previously diagnosed disease of respiratory, cardiovascular, endocrinology, liver, kidney, hematology, neurology and psychology function or other significant diseases and history
  * Known allergy or hypersensitivity to the study medication
  * AST or ALT greater than 1.25 times the upper limit of reference range or Total bilirubin greater than 1.25 times the upper limit of reference range base on screening results
  * A subject judged ineligible by the investigator to participate in this study for other reason containing clinical laboratory tests

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Safety
  Adverse events, Physical exam, Vital sign, Laboratory, 12-lead-ECG

SECONDARY OUTCOMES:
Pharmacokinetics
  AUC and Cmax in plasma